CLINICAL TRIAL: NCT00000419
Title: Safety of Estrogens in Lupus Erythematosus - National Assessment (SELENA): Hormone Replacement Therapy
Brief Title: Safety of Estrogens in Lupus: Hormone Replacement Therapy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Office of Research on Women's Health (ORWH) (NIH)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: U01 AR42540 NIAMS-028A; U01AR042540 (NIH)
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Systemic Lupus Erythematosus
Keywords: SLE; SELENA; Estrogen Replacement Therapy (ERT); Postmenopause; Osteoporosis; Estrogens; Steroids; Progestin; Placebo
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Osteoporosis | interventions — Estrogens, Conjugated (USP); Medroxyprogesterone Acetate

INTERVENTIONS:
Drug: Premarin and Provera

SUMMARY:
Safety of Estrogens in Lupus Erythematosus - National Assessment (SELENA) is a study to test whether postmenopausal women with systemic lupus erythematosus (SLE, or lupus) can safely use the hormone estrogen. In this part of the study, we will look at the effects of estrogen replacement therapy on the activity and severity of disease in women with SLE.

DETAILED DESCRIPTION:
This study tests the effect of exogenous female hormones on disease activity and severity in women with systemic lupus erythematosus (SLE). Physicians generally do not prescribe hormone replacement therapy (HRT) to women with SLE because of the widely held view that such treatment can activate SLE. This practice is based on the greater incidence of SLE in women than in men, biologic abnormalities of estrogen metabolism, murine models of lupus, several anecdotes of patients having disease flares while receiving exogenous hormones, and a single retrospective study in patients with preexisting renal disease. By contrast, recent retrospective studies suggest that the rate of flare is not significantly increased in patients taking HRT.

We will examine, in a multicenter, randomized, double-blind, placebo-controlled trial, the effect of hormonal replacement with conjugated estrogens on disease activity in postmenopausal women with SLE. We will recruit patients from clinics and private practices that include over 4,000 women with SLE, most belonging to minority groups.

We will give patients hormones for 1 year.

NOTE: This trial has been terminated as of August 2002 upon recommendation of the Data Safety Monitoring Board (DSMB), based on the findings of the WHI Trial. Study subjects have discontinued study drug but will continue followup visits to study doctors through May 2003

ELIGIBILITY:
Inclusion Criteria:

* Female
* Unequivocal diagnosis of SLE
* Inactive disease or stable on 0.5 mg/kg/day or less of prednisone
* Chemical evidence of menopause or have stopped periods for at least 6 months

Exclusion Criteria:

* Blood pressure >145/95 on three occasions
* Deep vein, arterial thrombosis or pulmonary embolus
* GPL >40; MPL >40; APL >50; dRVVT >37 sec
* APL antibody syndrome ever
* Gynecologic or breast cancer
* Hepatic dysfunction or liver tumors
* Diabetes mellitus (NOT due to steroids) with vascular disease
* Congenital hyperlipidemia
* Complicated migraine
* Severe disease activity (SLEDAI >12)
* Increase in SLEDAI >2 points in 3 months
* Unexplained vaginal bleeding
* Use of estrogen (HRT or OCP) for >1 month at any time after SLE diagnosis
* FSH <40
* Premenopausal myocardial infarction

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350
Dates: Start 1996-04; Study Completion 2002-08

CONTACTS AND LOCATIONS:
Overall Officials: Jill Buyon, M.D., Principal Investigator — Hospital for Joint Diseases, Department of Rheumatology; Michelle Petri, M.D., Study Director — Johns Hopkins Hospital, Department of Rheumatology
Locations (16):
- United States (16):
  - UAB Medical Center, Birmingham, Alabama
  - UCLA Medical Center, Dept. of Rheumatology, Los Angeles, California
  - University of Chicago Pritzker School of Medicine, Chicago, Illinois
  - Louisiana School of Medicine, Shreveport, Louisiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Univ. of Michigan Med. Ctr., Rheumatology Div., Ann Arbor, Michigan
  - Hospital for Joint Diseases, New York, New York
  - Hospital for Special Surgery, New York, New York
  - Albert Einstein College of Medicine, Jacoby Hospital, Dept. of Rheumatology, The Bronx, New York
  - UNC Medical Center, Dept. of Rheumatology, Chapel Hill, North Carolina
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Univ. of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Univ. of Pittsburgh, Dept. of Rheumatology, Pittsburgh, Pennsylvania
  - University of Texas Health Sciences Center, Houston, Texas
  - Medical College of Virginia, Ambulatory Care Center, Richmond, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Background] Petri M, Buyon J, Kim M. Classification and definition of major flares in SLE clinical trials. Lupus. 1999;8(8):685-91. doi: 10.1191/096120399680411281. PMID 10568907
- [Background] Kim MY, Buyon JP, Petri M, Skovron ML, Shore RE. Equivalence trials in SLE research: issues to consider. Lupus. 1999;8(8):620-6. doi: 10.1191/096120399680411308. PMID 10568898
- [Background] Buyon JP. Clinical trials in systemic lupus erythematosus. Curr Rheumatol Rep. 2000 Feb;2(1):11-12. doi: 10.1007/s11926-996-0062-y. No abstract available. PMID 11123033
- [Background] Buyon JP. Hormone replacement therapy in postmenopausal women with systemic lupus erythematosus. J Am Med Womens Assoc (1972). 1998 Winter;53(1):13-7. PMID 9458619
- [Background] Buyon JP, Dooley MA, Meyer WR, Petri M, Licciardi F. Recommendations for exogenous estrogen to prevent glucocorticoid-induced osteoporosis in premenopausal women with oligo- or amenorrhea: comment on the American College of Rheumatology recommendations for the prevention and treatment of glucocorticoid-induced osteoporosis. Arthritis Rheum. 1997 Aug;40(8):1548-9. doi: 10.1002/art.1780400831. No abstract available. PMID 9259444
- [Background] Buyon JP, Wallace DJ. The endocrine system, use of exogenous estrogens, and the urogenital tract. In Dubois' Lupus Erythematosus, 6th edition. Wallace DJ, Hahn BH, eds. Philadelphia: Lippincott Williams & Wilkins, 2002; pp. 821-841.
- [Result] Buyon JP, Petri MA, Kim MY, Kalunian KC, Grossman J, Hahn BH, Merrill JT, Sammaritano L, Lockshin M, Alarcon GS, Manzi S, Belmont HM, Askanase AD, Sigler L, Dooley MA, Von Feldt J, McCune WJ, Friedman A, Wachs J, Cronin M, Hearth-Holmes M, Tan M, Licciardi F. The effect of combined estrogen and progesterone hormone replacement therapy on disease activity in systemic lupus erythematosus: a randomized trial. Ann Intern Med. 2005 Jun 21;142(12 Pt 1):953-62. doi: 10.7326/0003-4819-142-12_part_1-200506210-00004. PMID 15968009